CLINICAL TRIAL: NCT06107712
Title: Does Onlıne Yoga Have Sımılar Effects Compared to Face-To-Face Yoga in Terms of Dıaphragm Thıckness, Body Balance and Psychosocıal Status?
Brief Title: Onlıne Yoga Compared to Face-To-Face Yoga on Dıaphragm Thıckness, Body Balance and Psychosocıal Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Bahar Ozgul, Assist Prof, PhD PT, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 25.06.2020/44
Record Dates: First submitted 2023-10-18; First posted 2023-10-30 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Mind-Body Therapies; Yoga; Telerehabilitation
Keywords: Yoga; Postural Balance; Telerehabilitation; Diaphragm; Ultrasonography; Mental Health; Pandemics
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online yoga exercise group (Experimental): Online yoga practice was implemented in a calm and quiet environment in the individuals' own home or dormitory in a way that they could participate online.
  Interventions: Other: Online yoga exercise
- Face-to-face yoga exercise group (Active Comparator): Face-to-face yoga practice was carried out at therapeutic exercise laboratory at Marmara University Health Sciences Faculty.
  Interventions: Other: Face-to-face yoga exercise
- control (No Intervention): Participants in the control group who continued their routine activities for six weeks after the initial evaluation and did not participate in any exercise, yoga, etc. program were included in the second evaluation.

INTERVENTIONS:
Other: Online yoga exercise — The basic yoga poses of Shivananda Yoga included in the online yoga group were shoulder stand (sarvangasana), plough pose (halasana), fish pose (matsyasana), backstretch (paschimothanasana), cobra (bhujangasana), locust (shalabhasana), bow (dhanurasana), spinal twist (matsyendrasana), crow pose (kakasana), standing backstretch (pada hasthasana) and triangle pose (trikonasana).
  The yoga practice flow was designed for individuals who had never practiced yoga before. In the initial classes, there was a focus on breathing exercises and warming-up series such as "Sun Salutations". The instructor frequently reminded the participants to perform all the poses with full yoga breaths and without holding their breath.
  In the scope of the study, the physiotherapist researcher who is a certified as the Shivananda Yoga instructor, performed the same yoga practice flow and steps in the both groups during six-week.
  Arms: Online yoga exercise group
Other: Face-to-face yoga exercise — The basic yoga poses of Shivananda Yoga included in the face-to-face yoga group were shoulder stand (sarvangasana), plough pose (halasana), fish pose (matsyasana), backstretch (paschimothanasana), cobra (bhujangasana), locust (shalabhasana), bow (dhanurasana), spinal twist (matsyendrasana), crow pose (kakasana), standing backstretch (pada hasthasana) and triangle pose (trikonasana).
  The yoga practice flow was designed for individuals who had never practiced yoga before. In the initial classes, there was a focus on breathing exercises and warming-up series such as "Sun Salutations". The instructor frequently reminded the participants to perform all the poses with full yoga breaths and without holding their breath.
  Arms: Face-to-face yoga exercise group

SUMMARY:
The goal of this randomized controlled study was to compared six-week online yoga program with six-week face-to-face yoga program on diaphragm thickness, body balance and physio social status in young female individuals. The main questions it aims to answer are:

* Does online yoga have similar effects compared to face-to-face yoga in terms of diaphragm thickness?
* Does online yoga have similar effects compared to face-to-face yoga in terms of body balance?
* Does online yoga have similar effects compared to face-to-face yoga in terms of psychosocial status such as level of anxiety and social media addiction? Participants completed the experimental steps of ultrasound scanning, balance testing and the scales questioning psychosocial status before and after 6-week online yoga program. After the pandemic conditions normalized, new participants were invited, and a 6-weeks face-to-face yoga program was applied and the same tests were applied before and after the program. As a control group, individuals whose physical activity levels were monitored and who did not participate in any exercise program were evaluated twice, six weeks apart. The researchers compared these three groups and examined whether there were differences between the groups in terms of the investigated parameters.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) has caused a major impact on physical activity behaviors worldwide due to the necessity of quarantine condition. Decreased physical activity due to isolation has the potential to worsen various health conditions, including various chronic diseases. Because of the positive effects of physical activity on the immune system during the COVID-19 epidemic, home-based tele-exercise programs have been considered a potential tool to maintain physical and mental health during the pandemic. During a period of inactive life, such as a pandemic, yoga exercises were among the home-based exercise programs for the general adult population. In addition to the effects of yoga on improvement of physical features such as respiratory capacity, muscle strength and balance, it is well known to have positive effects on supporting mental well-being and anxiety and stress levels.

Considering the literature, the effects of some physical exercise applications of home-based teleexercises, which started and as the continued during inactive life processes such pandemic period, were examined. However, no study has been found examining the effects of online yoga practice, especially on the basic respiratory muscle diaphragm structure and physical properties. Considering the physical and mental effects of yoga, the aim of this study was to evaluate the effect of yoga practice as teleexercise on psychosocial factors such as diaphragm muscle thickness, balance performance and anxiety, and social media addiction, compared to face-to-face practice, in a period where individuals have to spend a sedentary and inactive period due to the pandemic. It was thought that the results of the study will help to gain more detailed information about the effectiveness of teleexercise applications that continue to be implemented after the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-25 who were continuing their university education
* who had not practiced yoga regularly before
* who had not engaged in regular exercise for the last six months
* who had no psychosocial problems

Exclusion Criteria:

* Individuals who had undergone feet, knee, hip, or spine surgeries
* had musculoskeletal pain or neurological problems related to orthopaedic, cardiopulmonary, cardiovascular, or rheumatic diseases; pregnant
* had a body mass index over 30
* who did not participate in two or more yoga sessions

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic Ultrasonic Scanning | Baseline (T0, before beginning of the study); T1 (end of the 6-week programme/control period)
  Ultrasound scanning of the diaphragm was performed by a certificated physiotherapist. The researcher was blind to physical performance testing procedure and groups of participants.
  Real time ultrasound was performed to identify the intercostal space at which the diaphragm was most easily visualized between 2 ribs in the supine position. The eighth or ninth intercostal space at the anterior axillary line was imaged. When the ultrasound probe was located correctly to the intercostal space was identified, the subject was instructed to deep inhale and exhale slowly, and three images were collected at the point of maximum and minimum diaphragm thickness as identified visually by the examiner. The diaphragm was screened by its characteristic 3-layered appearance, location under the intercostal muscles and subcutaneous tissue. The thickness of diaphragm was frequently displayed thickest while inhaling at maximum level and thinnest while exhaling at maximum level.

SECONDARY OUTCOMES:
Body Balance Performance Testing | Baseline (T0, before beginning of the study); T1 (end of the 6-week programme/control period)
  The Balance Master device was used to perform limits of stability and weight bearing squat tests to assess motor status, and unilateral stance tests to assess functional limitations.
  The Limits of Stability: The subject was asked to keep the center of gravity on the central target by her/his postural control and perform the test by moving towards the target and remaining stationary on the target for eight seconds.
  The Weight Bearing(WBS)/Squat: The amount of body weight transferred to the feet was measured at four different degrees (0, 30, 60, 90) of knee flexion. The WBS symmetry score is expressed as a percentage by dividing the weight on one side by the total body weight. Good scores are those that are very close to 50% of body weight for each lower extremity.
  The Unilateral Stance: The test requires the participant to maintain balance on one foot while attempting to minimize postural sway with eyes open and closed for a duration of 10 seconds for each trial.

OTHER OUTCOMES:
Beck Depression Scale to detect level of distress | Baseline (T0, before beginning of the study); T1 (end of the 6-week programme/control period)
  Beck Depression Scale (BDS) is a self-evaluation scale consisting of 21 items scored between 0-3. The questions asked to the patient investigate how much the feeling of distress has bothered them in the past week. A high score indicates high levels of anxiety experienced by the individual.
Perceived Stress Scale to measure the degree of perceived stress | Baseline (T0, before beginning of the study); T1 (end of the 6-week programme/control period)
  The Perceived Stress Scale (PSS) is a 14-item questionnaire designed to measure the degree to which stress is perceived in various situations in a person's life. Each item is rated on a Likert-type scale ranging from never (0) to very often (4). A high score indicates high levels of perceived stress experienced by the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Zübeyir Sarı, Prof Dr, Study Director — Marmara University Health Science Faculty Physiotherapy and Rehabilitation Department; İlkşan Demirbüken, Prof Dr, Principal Investigator — Marmara University Health Science Faculty Physiotherapy and Rehabilitation Department; Leila Abdolalizadeh Khaselouei, PT, Principal Investigator — Marmara University Health Science Faculty Physiotherapy and Rehabilitation Department; Hilal B Can, MSc PT, Principal Investigator — Marmara University Health Science Faculty Physiotherapy and Rehabilitation Department; Mine G Polat, Prof Dr, Study Chair — Marmara University Health Science Faculty Physiotherapy and Rehabilitation Department; Bahar Özgül, PhD PT, Principal Investigator — Marmara University Health Science Faculty Physiotherapy and Rehabilitation Department
Locations (1):
- Bahar Özgül, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dor-Haim H, Katzburg S, Revach P, Levine H, Barak S. The impact of COVID-19 lockdown on physical activity and weight gain among active adult population in Israel: a cross-sectional study. BMC Public Health. 2021 Aug 6;21(1):1521. doi: 10.1186/s12889-021-11523-z. PMID 34362319
- [Background] Nieman DC, Wentz LM. The compelling link between physical activity and the body's defense system. J Sport Health Sci. 2019 May;8(3):201-217. doi: 10.1016/j.jshs.2018.09.009. Epub 2018 Nov 16. PMID 31193280
- [Background] Pecanha T, Goessler KF, Roschel H, Gualano B. Social isolation during the COVID-19 pandemic can increase physical inactivity and the global burden of cardiovascular disease. Am J Physiol Heart Circ Physiol. 2020 Jun 1;318(6):H1441-H1446. doi: 10.1152/ajpheart.00268.2020. Epub 2020 May 15. PMID 32412779
- See also: Organization, W. H. (2020). Coronavirus disease 2019 (COVID-19): situation report, 73 — https://www.who.int/publications/m/item/situation-report---73